CLINICAL TRIAL: NCT02108834
Title: Randomized Controlled Trial of Regional Anesthesia in Combination With General Anesthesia for Thyroidectomy
Brief Title: Regional Anesthesia for Thyroidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Principal Investigator, Xiangcai Ruan, Vice chair, Guangzhou First People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GZFPH-IRB-2013-085
Record Dates: First submitted 2014-04-04; First posted 2014-04-09 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Pain; Acute Pain
Keywords: chronic postsurgery pain; acute pain
MeSH Terms: conditions — Chronic Pain; Acute Pain | interventions — Nerve Block

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nerve block (Active Comparator): cervical plexus block with ropivacaine
  Interventions: Procedure: nerve block
- Placebo (Placebo Comparator): placebo saline
  Interventions: Procedure: placebo

INTERVENTIONS:
Procedure: nerve block — After general anaesthesia,the patient is placed in a supine position with the head turn away from the side to be blocked, and then the sternocleidomastoid muscle (SCM) is identified by slight head elevation. SCPB(superficial cervical plexus block) is performed with a 26-gauge needle that is inserted at the midpoint of the posterior border of the SCM muscle and the needle is advanced just past the SCM muscle. The mixture is prepared with 20ml of 0.5% ropivacaine in Group 1
  Arms: nerve block
Procedure: placebo — After general anaesthesia,the patient is placed in a supine position with the head turn away from the side to be blocked, and then the sternocleidomastoid muscle (SCM) is identified by slight head elevation. SCPB(superficial cervical plexus block) is performed with a 26-gauge needle that is inserted at the midpoint of the posterior border of the SCM muscle and the needle is advanced just past the SCM muscle. The mixture is prepared with 20ml of 0.9% saline in Group 2.
  Arms: Placebo

SUMMARY:
For more than 25 years, Regional Anesthesia has challenged anesthesiologists to determine whether it offers real benefits in terms of patient outcome from major surgery, compared with general anesthesia. Although it is clear that regional analgesia in association with general anesthesia substantially reduces postoperative pain, the benefits in terms of overall perioperative outcome are controversial. The aim of this study is to evaluate the effect on short and long-term postoperative outcomes of adding regional analgesia to general anaesthesia in thoridetomic patients.

DETAILED DESCRIPTION:
Patients who are divided into two treatment groups: (a) a bilateral superficial cervical plexus group (group S) and a control group (group C).We performe bilateral superficial cervical plexus block (BSCPB)with 0.25-0.75% ropivacaine10 ml to group S and 10ml NaCl 0.9% to group C. All BSCPB is performed by experienced anesthesia doctor after a standardized induction of general anaesthesia.eneral anaesthesia was induced by using intravenously with midazolam,propofol, fentanyl, cisatracurium is injected IV to facilitate orotracheal intubation. After a standardized induction of general anaesthesia, patients receive Regional Anesthesia at the discretion of the experienced anesthesiologist who was blinded to treatment.

The patient is placed in a supine position with the head turned away from the side to be blocked, and then the sternocleidomastoid muscle (SCM) is identified by slight head elevation. SCPB is performed with a 26-gauge needle that is inserted at the midpoint of the posterior border of the SCM muscle and the needle is advanced just past the SCM muscle.

ELIGIBILITY:
Inclusion Criteria:

-Eligible patients fit an ASA I or II classification adult patients who will be scheduled for elective thyroid lobectomy under general anaesthesia.

Exclusion Criteria:

* hypersensitivity to any study drugs
* Long-term use of anticoagulant drugs: warfarin or heparin
* the neck or systemic infection
* communication disorder
* refuse to accept this research subjects.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-02 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
the incidence of chronic postsurgery pain | 60 days
  the time from the end of surgery

SECONDARY OUTCOMES:
the intensity of acute pain | 24 hours
  swallowing pain and rest pain
hemodynamic stability | 1 day
  blood pressure and heart rate intraoperative responses.
postoperative nausea and vomiting | 2 days after operation

OTHER OUTCOMES:
The over-all satisfaction of patients | 24 hours
  The over-all satisfaction of patients after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xiangcai Ruan, MD, PHD, Principal Investigator — Guangzhou First Municipal People's Hospital,Guangzhou,Guangdong,China,510180
Locations (1):
- Guangzhou First Municipal People's Hospital, Guangzhou, China

REFERENCES:
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Dieudonne N, Gomola A, Bonnichon P, Ozier YM. Prevention of postoperative pain after thyroid surgery: a double-blind randomized study of bilateral superficial cervical plexus blocks. Anesth Analg. 2001 Jun;92(6):1538-42. doi: 10.1097/00000539-200106000-00038. PMID 11375842
- [Result] Brogly N, Wattier JM, Andrieu G, Peres D, Robin E, Kipnis E, Arnalsteen L, Thielemans B, Carnaille B, Pattou F, Vallet B, Lebuffe G. Gabapentin attenuates late but not early postoperative pain after thyroidectomy with superficial cervical plexus block. Anesth Analg. 2008 Nov;107(5):1720-5. doi: 10.1213/ane.0b013e318185cf73. PMID 18931238